CLINICAL TRIAL: NCT07382752
Title: Metabolomic and Genetic Factors Decoupling Immune Checkpoint Inhibitor Tumor Efficacy and Cardiovascular Toxicity
Brief Title: Decoupling Immunotherapy Toxicity and Cancer Response
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1571; NCI-2025-09341 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Tumor; Cardiovascular
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Observational Cohort: Utilizing baseline biospecimens for analysis of predictors of cardiotoxicity events and cancer outcomes after ICI initiation.

SUMMARY:
This study is a novel evaluation of cardiotoxicity after ICI therapy based on traditional CV risk factors with the addition of metabolomic profiles, epigenetic aging, and CHIP. It is not an extension of previous work in ICI therapy.

DETAILED DESCRIPTION:
Primary Objectives:

To identify predictors of a composite outcome comprising immune checkpoint inhibitor associated cardiovascular disease (ICI-CVD) and/or cancer progression or death.

To decouple the predictors of ICI-CVD and cancer treatment efficacy.

Secondary Objectives:

To identify human monocyte derived macrophages (HMDM)-derived metabolite signatures predictive of cardiovascular toxicity and cancer outcomes in ICI-treated patients.

To identify genetic (CHIP) and epigenetic age determinants of ICI-CVD and cancer outcomes in ICI-treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Plan to start immune checkpoint inhibitor for cancer therapy

Exclusion Criteria:

1. No baseline blood collection prior to initiation
2. At time of evaluation not determined to be a good candidate for evaluation of outcome events by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Palaskas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org